CLINICAL TRIAL: NCT07027930
Title: A Feasibility Trial of Eye Movement Desensitization and Reprocessing Therapy- Integrative Treatment Group Protocol for Ongoing Traumatic Stress in Road Traffic Accident Survivors for Reduction of Post-Traumatic Stress Symptoms
Acronym: EMDR-IGTP-OTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Punjab (Other)
Responsible Party: Principal Investigator, Khawer Javed, Principal Investigator, University of the Punjab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IGTP-OTS-MSCCP-2022
Record Dates: First submitted 2025-05-30; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Post Traumatic Stress Symptoms; Quality of Life (QOL); Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR-IGTP-OTS (Experimental): Eye movement desensitization and reprocessing therapy for ongoing traumatic stress
  Interventions: Other: Eye movement desensitization and reprocessing therapy integrative group treatment protocol for Ongoing traumatic stress
- Comparison Arm (No Intervention): This would be used as a control arm

INTERVENTIONS:
Other: Eye movement desensitization and reprocessing therapy integrative group treatment protocol for Ongoing traumatic stress — EMDR-IGTP-OTS is a group intervention based on EMDR 8-phased protocols with the integration of the Butterfly hug technique.
  Arms: EMDR-IGTP-OTS

SUMMARY:
Road traffic accidents (RTAs) are a significant public health concern globally, accounting for a substantial proportion of morbidity and mortality. This study evaluates the feasibility and acceptability of the Eye Movement Desensitization and Reprocessing Integrative Group Treatment Protocol for Ongoing Traumatic Stress (EMDR-IGTP-OTS) in the reduction of posttraumatic stress symptoms, depression, and anxiety, while improving the quality of life in individuals who have experienced traffic accidents. Using a randomized control design, participants aged 18-45 will be assessed at three-time points: pre-treatment, post-treatment, and one-month follow-up. The study employs the DASS-21, UIES-R, and WHOQOL-BREF as evaluation measures. Findings aim to expand evidence on trauma-focused interventions and explore their applicability in culturally diverse, resource-constrained settings.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years.
* Experienced a traffic accident 3 months to 10 years prior
* Willing to participate and able to understand the intervention components.

Exclusion Criteria:

* Participants will be excluded from the study if they meet any of the following criteria:

  * Diagnosed with conditions such as schizophrenia or bipolar disorder, which require specialized treatment beyond the scope of this study.
  * History of severe head injuries resulting in neurological or cognitive deficits.
  * Participants who have experienced a traffic accident less than 3 months ago, as immediate post-traumatic responses may not have stabilized

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The Urdu Impact of Event Scale-Revised | From Enrollment to end of study after 4 weeks
  It will measure trauma-specific symptoms such as intrusion, avoidance, and hyperarousal. This 22-item scale uses a 5-point Likert scale ranging from 0 (not at all) to 4 (extreme), comprehensively evaluating the psychological impact of traumatic incidents. Higher the scores, Higher will be severity of post traumatic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Khawer Javed, MS clinical Psychology, Principal Investigator — Centre for clinical Psychology, University of the Punjab
Locations (1):
- Public Universities, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to concerns regarding participant confidentiality, especially given the sensitive nature of trauma-related experiences addressed in the study. Although anonymization procedures are in place, the qualitative nature of the data and small sample size may still pose a risk of indirect identification. Therefore, to uphold ethical standards and protect participant privacy, we have decided not to share IPD publicly

REFERENCES:
- [Background] Yasar AB, Konuk E, Kavakci O, Uygun E, Gundogmus I, Taygar AS, Uludag E. A Randomized-Controlled Trial of EMDR Flash Technique on Traumatic Symptoms, Depression, Anxiety, Stress, and Life of Quality With Individuals Who Have Experienced a Traffic Accident. Front Psychol. 2022 Mar 24;13:845481. doi: 10.3389/fpsyg.2022.845481. eCollection 2022. PMID 35401305

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT07027930/Prot_SAP_ICF_000.pdf